CLINICAL TRIAL: NCT03658928
Title: Guangdong Association of Clinical Trials
Brief Title: A Non-interventional Retrospective Study on Overall Survival in Completely Resected Chinese NSCLC Patients With Adenocarcinoma Histology- ICAN Extension Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG1802
Record Dates: First submitted 2018-08-31; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-03

CONDITIONS: Overall Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ICAN was a non-interventional study to explore the EGFR gene mutation status, clinical outcome and recurrent risk factors in early stage Chinese NSCLC with adenocarcinoma histology after complete resection (NIS-OCN-DUM-2009/1). The study had enrolled 571 patients from Apr. 2010 to Dec. 2010 in 24 sites located in the mainland of China. The study had completed and major results showed that EGFR mutation rate was 55.1% and 3-year DFS rate was 61.7% in early stage Chinese NSCLC with adenocarcinoma histology after complete resection. Postoperative pathologic stage, gender, surgical and resection types had a statistically significant association with 3-year DFS.

This study is ICAN extension study with the purpose to collect the overall survival data from previous ICAN study. Approximately 571 patients who participated in ICAN study will be enrolled.

DETAILED DESCRIPTION:
Primary objective

* To observe the overall survival of early stage NSCLC with adenocarcinoma histology after complete resection that had enrolled in I CAN study.

Secondary objectives

* To observe the updated DFS of early stage NSCLC with adenocarcinoma histology after complete resection that had enrolled in I CAN study;
* To observe the treatment pattern after tumor recurrence of early stage NSCLC with adenocarcinoma histology after complete resection that had enrolled in I CAN study in real-world setting;
* To explore the risk factors of OS for early stage NSCLC with adenocarcinoma histology after complete resection that had enrolled in I CAN study in real-world setting, such as EGFR mutation status, gender, smoking history, treatment pattern after recurrence, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years old.
2. Provision of informed consent prior to any study specific procedures
3. Histological diagnosed as adenocarcinoma type of non-small cell lung cancer
4. Have completed lung cancer operation
5. The tumour EGFR gene mutation status test was performed as regular medical practice

Exclusion Criteria:

1. No provision of informed consent or EC approve informed consent waiver prior to any study specific procedures;
2. Patients withdrew consent for ICAN study;
3. Patients in whose medical record was objected to use the existing data for scientific research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is a non-interventional, retrospective study and all the patients participated in ICAN study will be enrolled.
Sampling Method: Probability Sample
Enrollment: 571 (Estimated)
Dates: Start 2018-08-31 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | from the date of operation to date of death from any cause, whichever came first, assessed up to 8 years.
  is defined as the time from the date of operation to date of death. For patients who are still alive, the last date when the patient is known to be alive will be used to determine the censoring date.

SECONDARY OUTCOMES:
Disease free survival | •from operation until recurrence of tumor or death from any cause, whichever came first, assessed up to 8 years.
  is defined as the time from operation until recurrence of tumor or death from any cause, whichever occurs first.